CLINICAL TRIAL: NCT05653336
Title: A Multicentre, Single-Arm, Pivotal Study to Evaluate the Safety and Efficacy of the Vivasure PerQseal® Closure Device System When Used to Achieve Haemostasis of Common Femoral Arteriotomies Created by 12 to 22 F Sheaths in Patients Undergoing Percutaneous Catheter-Based Interventional Procedures
Brief Title: PerQseal® Clinical Study
Acronym: PATCH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vivasure Medical Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P696-00
Record Dates: First submitted 2022-12-07; First posted 2022-12-16 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Percutaneous Large Hole Vascular Closure
Keywords: Vascular Closure; Vascular Closure Device; Large hole percutaneous closure; Large bore percutaneous closure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Subjects implanted with PerQseal Vascular Closure Device (Experimental): Subjects implanted with bioabsorbable implant to achieve haemostasis of common femoral arteriotomies created by 12 to 22 F sheaths (up to 26 F arteriotomy) in patients undergoing percutaneous catheter-based interventional procedures.
  Interventions: Device: PerQseal® Closure Device System

INTERVENTIONS:
Device: PerQseal® Closure Device System — Bioabsorbable implant delivered percutaneously to achieve haemostasis of common femoral arteriotomies created by 12 to 22 F sheaths (up to 26 F arteriotomy) in patients undergoing percutaneous catheter-based interventional procedures.

SUMMARY:
The objective is to evaluate the safety and effectiveness of the PerQseal vascular closure device system when used to achieve haemostasis of common femoral arteriotomies created by 12 to 22 F sheaths (arteriotomy up to 26 F) in subjects undergoing percutaneous catheter-based interventional procedures.

DETAILED DESCRIPTION:
The objective of this pivotal study is to evaluate the safety and effectiveness of the PerQseal vascular closure device system when used to achieve haemostasis of common femoral arteriotomies created by 12 to 22 F sheaths (arteriotomy up to 26 F) in subjects undergoing percutaneous catheter-based interventional procedures, with sufficient rigor to provide robust scientific evidence for the demonstration of clinical safety and efficacy of the PerQseal closure system to support a pre-market approval submission.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 19 years,
2. Clinically indicated for a percutaneous arterial interventional catheter-based procedure, e.g., transcatheter aortic valve replacement/implantation (TAVR/TAVI) or endovascular abdominal aortic aneurysm repair (EVAR), or thoracic endovascular aortic aneurysm repair (TEVAR), or use of a circulatory assist device or extracorporeal oxygenation using a common femoral arteriotomy created by a 12 to 22 F sheath (arteriotomy up to 26 F),
3. Subject is willing and able to provide appropriate study-specific informed consent, follow protocol procedures, and comply with follow-up visit requirements,
4. Females who are not pregnant or lactating and not planning to become pregnant for the duration of the study.

Baseline Exclusion Criteria:

1. Evidence of current systemic bacterial or cutaneous infection, including groin infection,
2. Known bleeding diathesis, definite or potential coagulopathy, platelet count < 100,000/µl or subjects on long term anticoagulants with an INR > 2 within 12 hours prior to index procedure,
3. Significant anaemia (haemoglobin < 9 g/dL or haematocrit < 27%), within 24 hours prior to index procedure,
4. Known type II heparin-induced thrombocytopenia,
5. Documented left ventricular ejection fraction < 20%,
6. Ipsilateral or contralateral lower extremity amputation.
7. Claudication (Rutherford category 3 or greater), documented untreated iliac or common femoral artery diameter stenosis > 50% or previous bypass surgery/stent placement in the common femoral artery of target leg,
8. Known existing nerve damage in the target leg,
9. Renal insufficiency (Glomerular Filtration Rate ≤ 30 ml/min or baseline serum creatinine > 2.5 mg/dL) or on renal replacement therapy,
10. Known allergy to any of the materials used in the PerQseal device (refer to Instructions for Use),
11. Subject unsuitable for surgical repair of the target leg access site,
12. Subject has undergone a percutaneous procedure greater than 8 F sheath in the target leg, within the 90-days prior to index procedure,
13. Subject has undergone a percutaneous procedure of 8 F sheath or less using an absorbable intravascular closure device for haemostasis, in the target leg, within the 90-days prior to index procedure,
14. Subject has undergone a percutaneous procedure of 8 F sheath or less using a suture mediated closure device or manual/mechanical pressure for haemostasis in the target leg, within the 30-days prior to index procedure,
15. Evidence of marked tortuosity of the femoral or external iliac arteries in the target leg, based on pre-primary procedure CT angiography,
16. Evidence of arterial diameter stenosis > 30% within 15 mm proximal or distal to arteriotomy site based on pre-primary procedure CT angiography,
17. Evidence of anterior wall calcification of the target common femoral artery (other than small, diffuse deposits which in the opinion of the investigator will not impede the vascular closure procedure) within 15 mm proximal or distal to arteriotomy site based on pre-primary procedure CT angiography,
18. Target femoral artery diameter is less than 6 mm or 7 mm, depending on whether S (small) or L (large) PerQseal Introducer will be used for arteriotomy closure, respectively, based on pre-primary procedure CT angiography,
19. Further planned endovascular/catheter-based procedure in the target leg in the 30-days following the index procedure.
20. Subject is enrolled in another investigational medical device or drug study,
21. Subject has been previously enrolled in this clinical study.
22. Current COVID-19 infection (with or without symptoms), recent positive test for COVID-19 within two weeks, or recent exposure to a person with COVID-19 infection within two weeks.

    Procedural Exclusion Criteria:

    If any Procedural Exclusion Criteria listed below are met, then closure with PerQseal device is not permitted.
23. Initial common femoral arterial access achieved with manual palpation or blind arterial stick access, without use of an image guided approach (ultrasound or angiography).
24. Difficult dilation during initial target femoral artery access (e.g., that damages or kinks dilators) while step-dilating up to the large-bore device,
25. During arterial puncture, the target femoral artery suspected to have experienced a posterior arterial wall needle puncture or underwent > one needle puncture during the primary procedure (with a needle larger than a Micropuncture needle (> 21 gauge or > 0.819 mm diameter) )
26. Subject has a tissue tract (i.e., estimated distance from skin entry point to arterial anterior surface at arteriotomy) expected to be greater than 8 cm.,
27. Significant blood loss requiring transfusion of blood products during primary procedure or within 30-days prior to index procedure,
28. Activated clotting time (ACT) > 250 seconds immediately prior to sheath removal or if ACT measurements are expected to be > 250 seconds for more than 24 hours after index procedure,
29. Target puncture site is in a vascular graft,
30. Target arteriotomy greater than 26 F,
31. Target arteriotomy in the profunda femoris or superficial femoral artery or is in common femoral artery, but within 15 mm proximal of the bifurcation of the superficial femoral/ profunda femoris artery,
32. Target arteriotomy located at the level or above the inferior epigastric artery and/or beneath or above the inguinal ligament based on bony/arterial landmarks (above femoral head on A-P projection),
33. Subjects with an acute haematoma > 4 cm diameter, arteriovenous fistula, pseudoaneurysm, or intraluminal thrombosis at the target access site identified intra-procedurally,
34. Evidence of bleeding around the primary procedure sheath (VARC type1/BARC type 2 or higher),
35. Intra-procedural angiographic evidence of arterial laceration, dissection or stenosis within the femoral artery that would preclude use of the PerQseal device,
36. Uncontrolled hypertension (systolic blood pressure > 180 mmHg or diastolic blood pressure > 110 mmHg) at the time of planned vascular closure,
37. Systolic blood pressure < 90 mmHg at the time of planned vascular closure.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint - Major Access Site Complications | through 30 days
  Rate of major access site complications attributable to the PerQseal device
Primary Effectiveness Endpoint - Time to Hemostasis | 20 Minutes
  Elapsed time in minutes from PerQseal (Introducer-sheath and Delivery Device) removal to first observed cessation of common femoral artery (CFA) bleeding, excluding cutaneous or subcutaneous oozing, and in the absence of a developing haematoma.

SECONDARY OUTCOMES:
Secondary Safety Endpoint - Minor Access Site Complications | through 30 Days
  Incidence of minor access site complications attributable to the PerQseal device
Secondary Effectiveness Endpoint - PerQseal Technical Success Rate | 10 Minutes
  Defined as the number of PerQseal devices that are deployed and achieve haemostasis (i.e., cessation of arterial bleeding excluding cutaneous or subcutaneous oozing) without need for more than 10 minutes of firm, adjunctive manual compression or alternative treatment (other than adjunctive endovascular ballooning) at target access site, divided by the total number of PerQseal devices where deployment was attempted. This is a per device endpoint.
Secondary Effectiveness Endpoint - PerQseal Treatment Success Rate | through 30 days
  Defined as the number of subjects who meet PerQseal Technical Success without experiencing a device related Major Access Site Complication through 30-days, divided by the total number of subjects where PerQseal device deployment was attempted.
Secondary Effectiveness Endpoint - Time to Device Deployment | 20 Minutes
  Defined as the time from insertion of the PerQseal delivery device into the PerQseal Introducer sheath to complete removal of the PerQseal (delivery device and introducer-sheath) from the subject following PerQseal deployment.
Secondary Effectiveness Endpoint - Time to Ambulation | through 24 hours
  Defined as the elapsed time from PerQseal removal until the subject can walk 20 feet/ 6 meters without arterial re-bleeding at the target access site. This endpoint will be evaluated only for subjects who are ambulatory (e.g., not confined to wheelchair or bed) at time of enrolment.
Secondary Effectiveness Endpoint - Total Closure Time | 40 Minutes
  Defined as time to Haemostasis plus Time to Device Deployment.

CONTACTS AND LOCATIONS:
Overall Officials: William Gray, Dr., Principal Investigator — Lankenau heart Institute; Sean Lyden, Dr., Principal Investigator — The Cleveland Clinic
Locations (18):
- United States (15):
  - HonorHealth, Scottsdale, Arizona
  - Scripps, La Jolla, California
  - Northern Light Eastern Maine Medical Center, Bangor, Maine
  - Cooper University Hospital, Camden, New Jersey
  - The Valley Hospital, Paramus, New Jersey
  - University of Buffalo, Buffalo, New York
  - Columbia University Medical Center/ NewYork Presbyterian Hospital, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Montefiore Medical Center (multiple centers), The Bronx, New York
  - The Cleveland Clinic, Cleveland, Ohio
  - UPMC Pinnacle Health, Mechanicsburg, Pennsylvania
  - UPenn - Perelman Center for Advanced Medicine,, Philadelphia, Pennsylvania
  - Lankenau Institute for Medical Research, Wynnewood, Pennsylvania
  - The Texas Heart Institute, Houston, Texas
- Germany (3):
  - St Franziskus Hospital, Münster, North Rhine-Westphalia
  - Leipzig University Hospital, Leipzig, Saxony
  - St. Gertrauden Krankenhaus (SGK), Berlin

IPD SHARING:
Plan to Share IPD: No